CLINICAL TRIAL: NCT00949663
Title: Xenin-25: Novel Regulator of Insulin Secretion and Beta-cell Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 08-0861B; 1R01DK088126-01 (NIH)
Record Dates: First submitted 2009-07-28; First posted 2009-07-30 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Blood Sugar; Xenin-25; GIP; Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance | interventions — Incretins; xenin 25

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Normal Glucose Tolerance (Experimental): Healthy individuals exhibiting plasma glucose levels less than 140mg/dl two hours after ingestion of 75-g of glucose.
  Interventions: Drug: Placebo; Drug: Glucose-dependent Insulinotropic Polypeptide (GIP); Drug: Xenin-25; Drug: Glucose-dependent Insulinotropic Polypeptide plus Xenin-25
- Impaired Glucose Tolerance (Experimental): Healthy individuals exhibiting plasma glucose levels between 140 and 199 mg/dl two hours after ingestion of 75-g of glucose.
  Interventions: Drug: Placebo; Drug: Glucose-dependent Insulinotropic Polypeptide (GIP); Drug: Xenin-25; Drug: Glucose-dependent Insulinotropic Polypeptide plus Xenin-25
- Type 2 Diabetes Mellitus (Experimental): Healthy individuals exhibiting plasma glucose levels greater than 150 mg/dL under fasting conditions OR greater than 199 mg/dl two hours after ingestion of 75-g of glucose.
  Interventions: Drug: Placebo; Drug: Glucose-dependent Insulinotropic Polypeptide (GIP); Drug: Xenin-25; Drug: Glucose-dependent Insulinotropic Polypeptide plus Xenin-25

INTERVENTIONS:
Drug: Placebo — Intravenous infusion of 1% human albumin in normal saline
  Other Names: Vehicle Alone
Drug: Glucose-dependent Insulinotropic Polypeptide (GIP) — Intravenous infusion of GIP (4 pmoles x kg-1 x min-1) in 1% human albumin in normal saline
  Other Names: GIP
Drug: Xenin-25 — Intravenous infusion of xenin-25 (4 pmoles x kg-1 x min-1) in 1% human albumin in normal saline
  Other Names: Xenin
Drug: Glucose-dependent Insulinotropic Polypeptide plus Xenin-25 — Intravenous infusion of GIP plus xenin-25 (4 pmoles each x kg-1 x min-1) in 1% human albumin in normal saline
  Other Names: GIP plus Xenin

SUMMARY:
An intestinal hormone called Glucose-dependent Insulinotropic Polypeptide (GIP) is released into the blood immediately after ingestion of a meal and plays an important role in regulating blood sugar levels. However, GIP is not active in persons with type 2 diabetes mellitus (T2DM) which is also known as adult onset or non-insulin-dependent diabetes. This study is being conducted to determine whether a hormone called xenin-25 can restore the activity of GIP in persons with T2DM.

DETAILED DESCRIPTION:
Each eligible participant will be administered an oral glucose tolerance test so he/she can be assigned to the group with "normal glucose tolerance", "impaired glucose tolerance" (between normal and diabetic), or type 2 diabetes mellitus. Each study subject will then be administered a meal tolerance test (MTT) on 4 separate occasions. For the MTT, a liquid meal (Boost Plus)will be ingested following an overnight fast. A primed-continuous infusion of vehicle alone, GIP alone, xenin-25 alone, or the combination of GIP plus xenin-25 (each peptide at a dose of 4 pmoles x kg-1 x min-1) will be initiated at the same time the meal is ingested. Blood samples will be collected before and during the MTT for the measurement of glucose, insulin, C-peptide, glucagon, GIP and xenin-25 levels.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65. No minors will be studied.
* Individuals must be able to consent for their own participation (no mental impairment affecting cognition or willingness to follow study instructions).
* Healthy volunteers with no clinical evidence of T2DM (see below).
* Otherwise healthy volunteers that have impaired glucose tolerance (see below).
* Otherwise healthy volunteers with Diet Controlled T2DM (see below).
* Otherwise healthy volunteers with T2DM that take oral agents only and if the subject's pre-existing oral anti-diabetic agents can be safely discontinued for 48 hours prior to Oral Glucose Tolerance Test.
* Otherwise healthy volunteers with T2DM who do not use insulin for blood glucose control.
* Persons with HbA1c ≤ 9%.
* Women of childbearing potential must be currently taking/using a method of birth control that is acceptable to the investigators. A pregnancy test will be done at the beginning of each visit. Any woman with a positive pregnancy test will be removed from the study.
* Willingness to return have 8-10ml of blood drawn 25-30 days after the last Xenin infusion; to check for Xenin peptide antibodies that MAY develop. (All efforts will be made to complete this visit during study participation.

Exclusion Criteria:

* <18years of age or >65 years of age
* Lacks cognitive ability to sign the consent &/or follow the study directions for themselves
* Women unwilling to comply with using an acceptable method of contraception during the course of the study, or who are currently breast-feeding.
* Any subject whose screening HbA1c is >9.0%
* Type 2 diabetes requiring the use of supplemental insulin @ home
* Volunteers with a history of Acute Pancreatitis
* Volunteer with a history of Chronic Pancreatitis and/or risk factors for chronic pancreatitis including hypertriglyceridemia (triglycerides >400mg/ml) hypercalcemia (blood calcium level >11.md/dl) and/or the presence of gallstones.
* Volunteers with a history of gastrointestinal disorders, particularly related to gastric motility/emptying such as gastric bypass, documented gastro-paresis in diabetic volunteers.
* Volunteers with a history of cancer. Exception: skin cancer.
* Diabetics that have the potential to have a low blood sugar without them being aware that their blood sugar is low (hypoglycemia unawareness).
* Known heart, kidney. liver or pancreatic disease requiring medications.
* Subjects unwilling to allow the use of their own blood or the human albumin in the preparation of the peptides.
* Unwillingness to allow blood glucose level adjustment (if needed) with IV insulin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The effects of GIP, xenin-25, or a combination of GIP plus xenin-25 on insulin secretion and blood glucose levels | 3 years

SECONDARY OUTCOMES:
We will develop an assay to measure the normal fasting and postprandial concentrations of endogenous xenin-25 and determine whether they are altered in T2DM. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Burton Wice, PhD, Principal Investigator — Washington University School of Medicine; Dominic Reeds, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Chowdhury S, Reeds DN, Crimmins DL, Patterson BW, Laciny E, Wang S, Tran HD, Griest TA, Rometo DA, Dunai J, Wallendorf MJ, Ladenson JH, Polonsky KS, Wice BM. Xenin-25 delays gastric emptying and reduces postprandial glucose levels in humans with and without type 2 diabetes. Am J Physiol Gastrointest Liver Physiol. 2014 Feb 15;306(4):G301-9. doi: 10.1152/ajpgi.00383.2013. Epub 2013 Dec 19. PMID 24356886